CLINICAL TRIAL: NCT07085481
Title: The Influence Of Bupivacaine Temperature On Subtenon Block Characteristics: A Prospective, Randomized, Controlled Trial
Brief Title: Effect of Warm Bupivacaine on Subtenon Block.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amany Hazem abdelmaksood EL-deeb, lecturer of anaesthesia and intensive care, faculty of medicine, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Warm Bupivacaine for eye block
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cataract
Keywords: sub tenon, bupivacaine, sensory block, temperature
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: A single investigator who will not be involved in the further study steps or data collection will assess the patients for eligibility, explain the study protocol and anesthetic technique, obtain written informed consent, open the sealed opaque envelopes containing group allocation, prepare all solutions for each block identical syringe, and handle the syringes during the injection process. The investigator who will perform the block will be blinded to group allocation and will be allowed to enter the operative room after preparation of the injection solution. In addition, the study subjects and the investigator who will collect the data will be blinded to the study group. To maintain blinding, the block administrator will wear gloves, and the solution will be administered within 40 seconds of preparation to minimize temperature perception.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operating room temperature bupivacaine (Experimental): patients will receive local anesthetic (5ml containing 5mg bupivacaine) that will be on a sterile shelf in the operating room at 23°C. The empty syringes and needles will be also on the same shelf before their use.
  Interventions: Drug: room temperature Bupivacaine
- Warm bupivacaine (Experimental): patients will receive local anesthetic (5ml containing 5mg bupivacaine) warmed to 37◦C for 20 minutes. The empty syringes and needles, in their packaging, will be held at the same temperature for at least 2 hours before initiating the block.
  Interventions: Drug: warm Bupivacaine

INTERVENTIONS:
Drug: room temperature Bupivacaine — bupivacaine will be on a sterile shelf in the operating room at 23°C. The empty syringes and needles will be also on the same shelf before their use.
  Other Names: Non-warmed bupivacaine
  Arms: Operating room temperature bupivacaine
Drug: warm Bupivacaine — bupivacaine will be warmed to 37◦C for 20 minutes. The empty syringes and needles, in their packaging, will be held at the same temperature for at least 2 hours before initiating the block.
  Other Names: Pre-heated bupivacaine
  Arms: Warm bupivacaine

SUMMARY:
Sub-Tenon's anesthesia is now widely regarded as a preferred local anesthetic method for cataract surgery. Various techniques have been explored to prolong the duration, shorten onset time and improve the efficacy of local anesthetic nerve blocks with varying degrees of success. Warming local anesthetic may speed up its onset and prolong its effect by lowering its pKa.The aim of this study is to evaluate the effect of warming bupivacaine on the characteristics of a sub-Tenon's block in patients undergoing cataract surgery. It is hypothesized that warming bupivacaine 0.5% to 37°C will improve the characteristics of sub-Tenon's block. It will prolong the duration of sensory and motor block and accelerate the time onset time of sensory and motor block.

DETAILED DESCRIPTION:
Most ophthalmic surgeries are now conducted as day-case procedures under local anesthesia, which has improved efficiency, lowered costs, and enhanced safety, all while ensuring high levels of patient satisfaction. In cataract surgery, local anesthesia is widely favored, as it avoids the risks linked to general anesthesia. Sub-Tenon's anesthesia is now widely regarded as a preferred local anesthetic method for various ophthalmic procedures, especially cataract surgery. Compared to needle-based techniques, it presents several advantages, such as a reduced risk of globe injury, and increased safety for patients taking anticoagulant medications. Nonetheless, minor side effects like chemosis and subconjunctival hemorrhage remain common. When local anesthetic (LA) is delivered into the posterior sub-Tenon's space, it forms a fluid reservoir around the back of the globe, effectively blocking the ciliary nerves and providing anesthesia. Within 3-5 minutes, the anesthetic spreads along the sheaths of the extraocular muscles, diffuses into the intraconal space, and extends to the fascial planes around the eyelids, resulting in akinesia of the globe and orbicularis oculi muscle.The superior oblique muscle is typically the last to become akinetic, likely due to its distance from the globe and the fact that the trochlear nerve lies outside the muscle cone. The volume of LA used for Sub-Tenon's block varies among practitioners, typically ranging from 1 to 10 ml, with most using 2 to 5 ml. Smaller volumes can provide adequate anesthesia but may result in limited akinesia, while larger volumes offer quicker and more complete akinesia but increase the risk of chemosis and elevated intraocular pressure. Various LA agents, including lignocaine, bupivacaine and ropivacaine, have been used, either alone or in combination. A mixture of lignocaine 2% and bupivacaine 0.5% combines the advantages of a rapid block onset by lignocaine and longer effect and postoperative analgesia by bupivacaine, and it is popular among some anesthetists. Adding hyaluronidase can increase membrane permeability, improve the onset and quality of the block and reduce the median effective LA volume needed. A significant constraint of single-shot local anesthetic in the management of peri-operative analgesia is the limited duration of the nerve block. Liposomal bupivacaine was developed to circumvent this, but the duration of action remains controversial, it is expensive and not available in all countries. Various techniques have been explored to prolong the duration, shorten onset time and improve the efficacy of local anesthetic nerve blocks with varying degrees of success. Some of these involve mixing local anesthetics or adding adjuncts.Warming local anesthetic may speed up its onset and prolong its effect by lowering its pKa, thereby increasing the non-ionized fraction responsible for its pharmacological action. This approach has been studied in various regional blocks. However, there is limited research specifically examining the impact of warmed anesthetic on injection pain during ophthalmic blocks.

The aim of this study:

evaluate the effect of warming bupivacaine on the characteristics of a sub-Tenon's block in patients undergoing cataract surgery.

Sample Size Calculation:

Sample size was calculated using Power Analysis and Sample Size software program (PASS) version 3.1.9.2 for windows (2017). The primary outcome will be time to onset of sensory block. In a pilot study performed on 10 patients using room temperature bupivacaine, the mean (SD) of time to onset of sensory block was 8(3) minutes. Using a two-sided hypothesis test with a significance level of 0.05, assuming alpha = 0.05 and beta = 0.2 (power = 80%) and using a student t test, 57 subjects will be required in each group to detect 20 % difference between groups which is considered the minimal clinically important difference. To allow for subject dropouts, 60 subjects will be assigned to each group.

The study will be conducted in Mansoura ophthalmology center including 120 patients who will be scheduled for cataract surgery under local anesthesia. eligible patients will be randomly assigned to 2 equal groups (operating room temperature group) and (warm temperature group) according to computer-generated table of random numbers. The group allocation will be concealed in sequentially numbered, sealed opaque envelopes which will be opened only after obtaining the written informed consent.

All patients will be kept fasting according to pre-operative ASA recommendations prior to surgery. Basic demographic characters including age, gender, and BMI will be recorded.

The peri-operative management will be identical in both groups. All patients with planned day case cataract surgery under sub-Tenon's anesthesia will be assessed preoperatively by detailed medical history taking and physical examination. Investigations will be requested as appropriate. The 11-point NRS score (0 = no pain and 10 = the worst possible pain) will be explained to each patient.

On arrival to the anesthetic room, standard monitoring including 3 leads electrocardiogram (ECG), pulse oximetry, and noninvasive blood pressure will be applied. Baseline vital signs (heart rate and mean arterial blood pressure) will be recorded. Intravenous access will be established, and all patients will receive a single dose of prophylactic antibiotic after sensitivity test. No sedation will be administered A standardized sub-Tenon's block will be employed by the same consultant anesthetist to all patients within the study. The surface of the eye will be cleaned with two drops of 5% povidine iodine. The eyelids and orbital rim will be cleaned with 10% povidine iodine and an eye speculum will be inserted. A small incision will be made 5 mm from the limbus in the inferior-nasal quadrant. Blunt dissection will be used to identify the sub-Tenon's space. Once identified, a 19-G sub-Tenon's needle will be inserted, and the local anesthetic solution will be given slowly over 20 s. At no point during the administration of the injection the barrel of the syringe will be handled by consultant anesthetist.

Statistical Methods:

The collected data will be coded, processed, and analyzed using SPSS program (version 22) for Windows. Normality of numerical data distribution will be tested by Shapiro-Wilk test. Continuous data of normal distribution will be presented as mean ± SD and will be compared with the unpaired student's t test. Non-normally distributed data will be presented as median (range) and will be compared with the Mann-Whitney U test. Categorical data will be presented as number (percentage) and will be compared with the Chi-square test. All data will be considered statistically significant if P value is ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) I, II or III patients.
* Patients scheduled for elective unilateral cataract surgery.

Exclusion Criteria:

* Patient refusal to participate in the study.
* Altered mental status or un-cooperative patients or psychiatric disorder.
* History of anesthetic drug allergy.
* Pre-existing progressive demyelinating neurologic pathology or neuromuscular disorders.
* Any contraindications to block (as bleeding or coagulation diathesis).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
the time to onset of sensory block | Sensory blockade will be evaluated at 1, 2, 4, 6, 8, 10 and 15 minutes after injection, and then every 30 minutes after the end of surgery for 6 hours and end of block duration is defined by return of sensation.
  Sensory block (loss of sensation in the conjunctiva and sclera and indirectly optic nerve block) will be evaluated by touch the conjunctiva using cotton wisp or forceps in the inferior fornix and ask patient if they feel it, on a 3-point scale 0= No sensation (complete block) 1= reduction in sensation 2= on loss of sensation (no block), with identical contralateral testing as reference. Ask about vision or light perception; if the optic nerve is partially blocked, the patient may report blurred or lost vision- full optic nerve block causes temporary vision loss. The time to sensory block onset (the time elapsed from the end of injection and start of the loss of sensation score =1)

SECONDARY OUTCOMES:
time to complete sensory block | Sensory blockade will be evaluated at 1, 2, 4, 6, 8, 10 and 15 minutes after injection, and then every 30 minutes after the end of surgery for 6 hours and end of block duration is defined by return of sensation
  Sensory block (loss of sensation in the conjunctiva and sclera and indirectly optic nerve block) will be evaluated by touch the conjunctiva using cotton wisp or forceps in the inferior fornix and ask patient if they feel it, on a 3-point scale 0= No sensation (complete block) 1= reduction in sensation 2= on loss of sensation (no block), with identical contralateral testing as reference. Ask about vision or light perception; if the optic nerve is partially blocked, the patient may report blurred or lost vision- full optic nerve block causes temporary vision loss. time to complete sensory block(score = 0),
duration of sensory block | Sensory blockade will be evaluated at 1, 2, 4, 6, 8, 10 and 15 minutes after injection, and then every 30 minutes after the end of surgery for 6 hours and end of block duration is defined by return of sensation
  Sensory block (loss of sensation in the conjunctiva and sclera and indirectly optic nerve block) will be evaluated by touch the conjunctiva using cotton wisp or forceps in the inferior fornix and ask patient if they feel it, on a 3-point scale 0= No sensation (complete block) 1= reduction in sensation 2= on loss of sensation (no block), with identical contralateral testing as reference. Ask about vision or light perception; if the optic nerve is partially blocked, the patient may report blurred or lost vision- full optic nerve block causes temporary vision loss. duration of sensory block (defined as the elapsed time between the end of injection and the complete resolution and recovery to a normal sensory function)
The time to motor block onset | motor blockade will be evaluated at 1, 2, 4, 6, 8, 10 and 15 minutes after injection, and then every 30 minutes after the end of surgery for 6 hours
  Motor block (ocular akinesia) will be assessed by asking the patient to move the eye in the four cardinal directions; up ( superior rectus), down (inferior rectus), medially(medial rectus) , and laterally (lateral rectus) using Brahma score (0-3 for each direction) 0= No movement ( complete block) 1= marked reduction in movement 2= slight reduction in movement 3= full movement (no block), total maximum score= 12.The time to motor block onset (score = 8)
time to complete motor block | motor blockade will be evaluated at 1, 2, 4, 6, 8, 10 and 15 minutes after injection, and then every 30 minutes after the end of surgery for 6 hours
  Motor block (ocular akinesia) will be assessed by asking the patient to move the eye in the four cardinal directions; up ( superior rectus), down (inferior rectus), medially(medial rectus) , and laterally (lateral rectus) using Brahma score (0-3 for each direction) 0= No movement ( complete block) 1= marked reduction in movement 2= slight reduction in movement 3= full movement (no block), total maximum score= 12.time to complete motor block (score=0)
duration of motor block | motor blockade will be evaluated at 1, 2, 4, 6, 8, 10 and 15 minutes after injection, and then every 30 minutes after the end of surgery for 6 hours
  Motor block (ocular akinesia) will be assessed by asking the patient to move the eye in the four cardinal directions; up ( superior rectus), down (inferior rectus), medially(medial rectus) , and laterally (lateral rectus) using Brahma score (0-3 for each direction) 0= No movement ( complete block) 1= marked reduction in movement 2= slight reduction in movement 3= full movement (no block), total maximum score= 12.duration of motor block (defined as the elapsed time between the end of injection and the complete resolution of motor block)
Pain during injection | during injection only
  Pain during injection will be assessed using the 11-point NRS score (0 = no pain and 10 = the worst possible pain).
Patient satisfaction | before discharge only
  using a 4-point scale (1 = excellent,2= good, 3 = fair and 4 = poor).
surgeon satisfaction | at the end of the surgery
  using a 4-point scale (1 = excellent,2= good, 3 = fair and 4 = poor).
Incidence of adverse effects | Up to 6 hours after the procedure
  hypotension and bradycardia

CONTACTS AND LOCATIONS:
Overall Officials: Amany H ELDeeb, MD, Principal Investigator — Faculty of Medicine, Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The effect of warming ropivacaine on ultrasound-guided subgluteal sciatic nerve block: a randomized controlled trial — https://pmc.ncbi.nlm.nih.gov/articles/PMC10641952/
- See also: The Influence of Bupivacaine Temperature on Supraclavicular Plexus Block Characteristics: A Randomized, Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/?term=El+Bendary+HM&cauthor_id=33185376
- See also: The effect of warming ropivacaine on ultrasound-guided subgluteal sciatic nerve block: a randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/?term=Zhang+F&cauthor_id=37957544
- See also: Effect of temperature and pH adjustment of bupivacaine for intradermal anesthesia — https://pubmed.ncbi.nlm.nih.gov/?term=Jones+JS&cauthor_id=9517682